CLINICAL TRIAL: NCT03252730
Title: In-Use Test With a Cosmetic Product (WO 4260) for Topical Use on the Scalp
Brief Title: In-Use Test With a Cosmetic Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. August Wolff GmbH & Co. KG Arzneimittel (Industry)
Collaborators: SIT Skin Investigation and Technology Hamburg GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPT-15/2016
Record Dates: First submitted 2017-07-18; First posted 2017-08-17 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Dermatitis, Atopic
Keywords: Dry scalp; Itchy scalp
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WO 4260 Cosmetic Product for Topical Use (Experimental): WO 4260 is used to treat dry and itchy scalp
  Interventions: Other: WO 4260 Cosmetic Product for Topical Use

INTERVENTIONS:
Other: WO 4260 Cosmetic Product for Topical Use — Application on the hair scalp at least once a day over four weeks

SUMMARY:
The aim of the study is to evaluate the tolerance of the product WO 4260 by a dermatologist. Additional objectives of this clinical in-use study are to evaluate the cosmetic features and acceptance of the product by means of a questionnaire in an interview situation and by skin hydration measurements on the scalp.

ELIGIBILITY:
Inclusion Criteria:

* age: ≥ 18 years
* sex: approx. 50% male and approx. 50% female
* users of hair tonic for dry scalp
* dry, itchy scalp prone to atopic eczema / atopic dermatitis

Exclusion Criteria:

* any deviation from the above-mentioned criteria
* users of sour hair rinse
* subjects who wash their hair more than once a day
* other dermatological disorders (scars, moles) on the scalp
* known incompatibilities to cosmetics and ingredients of cosmetic test products (please see INCI)
* topical medication in the test area within 1 month prior to study start
* systemic medication with anti-inflammatory agents and antibiotics within 2 weeks prior to starting of the study
* systemic medication with retinoids, antihistamines and/or immunomodulators (e.g. cortisone, corticosterone, chemotherapeutic agents) within 4 weeks prior to starting of the study
* systemic illness of the subject at the beginning of the study
* pregnancy and period of breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
Tolerance of the Test Product on the Scalp | after 4 weeks of treatment
  Change from Baseline Tolerance on the Scalp at 4 weeks

SECONDARY OUTCOMES:
Skin Hydration of the Scalp | before product treatment; after 2 and 4 weeks of treatment
  The measurement is performed using the DermaLab® device with the moisture pin (Cortex Technology)
Performance of the Test Product | after 4 weeks of treatment
  Subjective assessment of product performance in a questionnaire-based interview
Tolerance of the Test Product on the Scalp | after 2 weeks of treatment
  Dermatological assessment of the Scalp concerning the Tolerance of the Test Product regarding erythema, edema dryness etc. Each item is scored 0=absent to 4=extreme.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Mazinani, MD, Study Director — SIT Skin Investigation and Technology Hamburg GmbH
Locations (1):
- SIT Skin Investigation and Technology Hamburg GmbH, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No